CLINICAL TRIAL: NCT02674789
Title: Ionized Magnesium Concentration in Athletes and Exercise Induced Changes in Ionized Magnesium
Brief Title: Ionized Magnesium in Athletes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Wageningen University (Other)
Collaborators: Gelderse Vallei Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: NL54333.081.15
Record Dates: First submitted 2015-12-09; First posted 2016-02-04 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-02

CONDITIONS: Magnesium Deficiency
Keywords: Exercise; Athletes; Ionized Magnesium; Variation; Blood
MeSH Terms: conditions — Magnesium Deficiency; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise day (Experimental): Behavioral intervention: 90min bike ergometer test at 70% of VO2max. Blood samples are collected at set time points (08:30, 11:00, 12:30, 13:30, 15:00, 16:00 and 18:30). Blood samples are analyzed on the pHOx analyzer for their ionized magnesium concentration. And on the Dimension Vista 1500 from Siemens for their total magnesium concentration.
  Interventions: Behavioral: Exercise protocol
- Non exercise day (Rest day) (No Intervention): No exercise protocol. Estimating daily variation of magnesium concentration. Blood samples are collected at set time points (08:30, 11:00, 12:30, 13:30, 15:00, 16:00 and 18:30). Blood samples are analyzed on the pHOx analyzer for their ionized magnesium concentration. And on the Dimension Vista 1500 from Siemens for their total magnesium concentration.

INTERVENTIONS:
Behavioral: Exercise protocol — 70% VO2max bike ergometer test for 90 minutes
  Arms: Exercise day

SUMMARY:
Ionized magnesium variation is measured during a normal day and again during a day with an exercise protocol of 90 minutes.

DETAILED DESCRIPTION:
Magnesium is an essential micronutrient for health and exercise performance. Deficiencies are common, especially in case of insufficient diets. Athletes are a population at risk of magnesium deficiency, as they can have strong nutritional (dis)believes and increased losses through sweat. That is why monitoring magnesium status in athletes is very important. Ionized magnesium is the active form of total magnesium, this value might be even more important than total magnesium. However, whether ionized magnesium is influenced by day variation is not clear yet. In addition: one bout of exercise can change magnesium status and probably ionized magnesium status. For people active in sports it is important to be aware of this variation in magnesium status, to prevent the diagnosis of false inadequate magnesium status. Therefore it is the aim of this proposal to determine whether ionized magnesium varies within one day and whether it changes after an acute bout of exercise.

Objective:

The main objective is to investigate whether ionized magnesium concentration varies during one day, and whether it is changed after one bout of exercise

Study design:

This will be a cross-over design. With screening and preliminary tests before the exercise test day and the non-exercise test day. The order in which exercise day and non-exercise day will be done, will be randomly divided between the participants.

Intervention:

A rest day and an exercise day At exercise day: an exercise test of 90 min at 70% of VO2max. Blood samples are taken at set time points during rest day and exercise day

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 - 45 y
* BMI: 18.5 - 25
* Minimal of 5 hours of training per week, for at least 2 years
* Used to bike, at least 5 hours per week in high season
* No Mg and / or Ca supplementation during study
* No blood donation, during or in the 6 weeks preliminary the study
* Suitable veins
* No chronic medication, with the exception of paracetamol and or birth control
* No antibiotics in the month preliminary the study
* Good health
* Serum Mg > 0.7 mmol/L
* Willing to give blood
* Able to be present and participate at all test days

Exclusion Criteria:

* Chronical illness
* Use of medication with the exception of paracetamol and or birth control
* Mg and or Ca supplementation use
* Inadequate Mg intake (according to FFQ)
* Working at Human Nutrition
* Wageningen University Msc thesis or internship at Human Nutrition
* Participating in other scientific research (with the exception of EetMeetWeet)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2015-12; Primary Completion 2016-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Blood samples analyzed on the pHOx analyzer for their ionized magnesium concentration | Blood samples are collected at 7 set time points during one day
  blood

SECONDARY OUTCOMES:
blood samples are analyzed on the Dimension Vista 1500 of Siemens for their total magnesium concentration | Blood samples are collected at 7 set time points during one day
  blood plasma

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Klein Gunnewiek, Phd, Principal Investigator — Gelderse Vallei Hospital

IPD SHARING:
Plan to Share IPD: Yes
Participants receive a letter with their personal information. VO2max, body weight and height, total Magnesium and ionized magnesium will be communicated.